CLINICAL TRIAL: NCT04768322
Title: Left Ventricular Assist Device (LVAD) Versus Guideline Recommended Medical Therapy in Ambulatory Advanced Heart Failure Patients (GDMT)
Brief Title: LVAD Versus GDMT in Ambulatory Advanced Heart Failure Patients
Acronym: AMBU-VAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL20_0072; ID-RCB (Other: 2020-A03451-38)
Record Dates: First submitted 2021-02-17; First posted 2021-02-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: End-stage Heart Failure
Keywords: Heart Failure; End-stage; Not inotrope-dependent; Left Ventricular Assist Device; HeartMate 3 system; Heart Surgery; Guideline Directed Medical Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Left Ventricular Assist Device and Guideline Directed Medical Therapy (Experimental): The intervention group will receive an early left ventricular assist device implantation (bridge to transplantation, bridge to candidacy or destination therapy) in addition to guideline directed medical therapy within 21 days of randomization.
  Interventions: Device: HeartMate 3 TM Left Ventricular Assist System; Other: Guideline Directed Medical Therapy
- Guideline Directed Medical Therapy (Other): Patients randomized in the control group will continue their guideline directed medical therapy which comprises the following stable combination at the maximal tolerated dose of betablockers, Angiotensin-Converting-Enzyme-inhibitors or Angiotensin II Receptor Blockers or Angiotensin receptor Neprilysin inhibitor and Mineralocorticoid Receptor Antagonists and Sodium-GLucose co-Transporter-2 (SGLT2) inhibitors if tolerated.
  Interventions: Other: Guideline Directed Medical Therapy

INTERVENTIONS:
Device: HeartMate 3 TM Left Ventricular Assist System — The HeartMate 3 TM Left Ventricular Assist System will be implanted within 21 days of randomization.
  Arms: Early Left Ventricular Assist Device and Guideline Directed Medical Therapy
Other: Guideline Directed Medical Therapy — Patients randomized in the control group will continue their guideline directed medical therapy which comprises the following stable combination at the maximal tolerated dose of betablockers, Angiotensin-Converting-Enzyme-inhibitors or Angiotensin II Receptor Blockers or Angiotensin receptor Neprilysin inhibitor and Mineralocorticoid Receptor Antagonists and Sodium-GLucose co-Transporter-2 (SGLT2) inhibitors if tolerated.

SUMMARY:
Heart failure is a severe disease affecting approximately 1-2% of the adult population in developed countries and around 26 million people worldwide. Up to 10% of these patients are in advanced stage heart failure, which is defined by a significant morbimortality and considerable medical expenses. Despite advances in its medical management, advanced (or end stage) heart failure is characterized by refractoriness to conventional therapies including guideline-directed pharmacological and non-surgical device treatments. These patients remain severely symptomatic (NYHA IV) and have objective signs of congestion or low cardiac output.

Left ventricular assist devices (LVADs) have been used in patients with heart failure with reduced ejection fraction for almost 20 years either as an alternative or a bridge to heart transplantation. LVADs improve heart failure symptoms and survival at the cost of increased rates of infection, stroke and bleeding.

Despite the lack of evidence, LVAD implantation in ambulatory patients is not rare, with INTERMACS profiles ≥4 patients representing 15.7% of the overall population implanted between 2012 and 2016.

The aim of this study is to investigate the efficacy and safety of left ventricular assist devices compared to traditional HF medical treatment alone in a population of ambulatory advanced heart failure patients. Secondary objectives are to better identify subgroups of patients that would benefit the most from the implantation of an LVAD as well as to assess the optimal timing of intervention.

ELIGIBILITY:
Inclusion Criteria:

1. All patients ≥18 years,
2. End-stage heart failure, evaluated by the local Heart Team, defined as:

   * Left ventricular ejection fraction ≤ 35% within 1 week prior to randomization and
   * Cardiac Index < 2.2 L/min/m² by hemodynamic use within 1 month prior to randomization or VO2 max < 14 ml/kg/min (or <50% of predicted VO2max) within 1 month prior to randomization OR low 6-min walking test (< 420 m) within 1 month prior to randomization or ≥ 2 hospitalizations for heart failure in the past year and
   * NYHA III-IV (INTERMACS profile 4-6) and and
   * Receiving medical management with optimal doses of betablockers, Angiotensin-Converting-Enzyme-inhibitors or Angiotensin II Receptor Blockers or angiotensin receptor neprilysin inhibitor (if eligible) and Mineralocorticoid Receptor Antagonists and Sodium-GLucose co-Transporter-2 (SGLT2) inhibitors for at least 45 days if tolerated according to guideline at maximal tolerated dose (if maximal HF drug dosage is not reached the investigators will have to explain reason behind not maximal dosage).
   * Receiving Cardiac Resynchronization Therapy and or Implantable Cardioverter Defibrillators if indicated for at least 45 days and
   * No mechanical circulatory support or inotrope therapy since > 30 days,
3. Having a health coverage,
4. Signed written informed consent,
5. Patient without any legal protection measure.

Exclusion Criteria:

1. Inotrope dependent patients or existence of ongoing mechanical circulatory support (MCS) in the last 30 days,
2. Right ventricular dysfunction (heart team consensus) with the expected need of Bi-VAD support,
3. Female patients currently pregnant or women of childbearing age who were not using contraception,
4. Active infection,
5. Irreversible end-organ dysfunction prior to LVAD implantation,
6. Contraindication to anti-coagulant or anti-platelet therapies,
7. History of any organ transplant prior to inclusion,
8. Psychiatric disease/disorder, irreversible cognitive dysfunction or psychosocial issues likely to impair compliance,
9. Frailty according to heart team,
10. Platelet count < 100,000 x 103/liter (<100,000/ml)
11. Body Surface Area (BSA) < 1.2 m2,
12. Any condition other than heart failure that could limit survival to less than 24 months,
13. Chronic renal insufficiency (GFR definitely <30 ml/min) or hepatic cirrhosis,
14. Participation in any other interventional clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality rate | Through 24 months when the last subject completes 12 months of follow-up
  The composite of 5 clinical endpoints is using a win ratio concept. Mortality has higher priority than Urgent ECMO implantation, urgent heart transplantation or LVAD implantation, unplanned hospitalization for heart failure, improvement of KCCQ by at least 5points, improvement of 6-minute walk test distance by at least 75 meters. Our main approach uses matched pairs of patients. Each pair is 'untied' first on the basis of the most important event (death) and secondly (if necessary) on the lesser event. The numbers of pairs in which the patient on new treatment 'won' and 'lost' are compared to produce the 'win ratio'. The 95% CI and P-value for the win ratio are readily obtained.
Number of urgent ECMO implantation | Through 24 months when the last subject completes 12 months of follow-up
  The composite of 5 clinical endpoints is using a win ratio concept. Mortality has higher priority than Urgent ECMO implantation, urgent heart transplantation or LVAD implantation, unplanned hospitalization for heart failure, improvement of KCCQ by at least 5points, improvement of 6-minute walk test distance by at least 75 meters. Our main approach uses matched pairs of patients. Each pair is 'untied' first on the basis of the most important event (death) and secondly (if necessary) on the lesser event. The numbers of pairs in which the patient on new treatment 'won' and 'lost' are compared to produce the 'win ratio'. The 95% CI and P-value for the win ratio are readily obtained.
Number of urgent heart transplantation | Through 24 months when the last subject completes 12 months of follow-up
  The composite of 5 clinical endpoints is using a win ratio concept. Mortality has higher priority than Urgent ECMO implantation, urgent heart transplantation or LVAD implantation, unplanned hospitalization for heart failure, improvement of KCCQ by at least 5points, improvement of 6-minute walk test distance by at least 75 meters. Our main approach uses matched pairs of patients. Each pair is 'untied' first on the basis of the most important event (death) and secondly (if necessary) on the lesser event. The numbers of pairs in which the patient on new treatment 'won' and 'lost' are compared to produce the 'win ratio'. The 95% CI and P-value for the win ratio are readily obtained.
Number of LVAD implantation | Through 24 months when the last subject completes 12 months of follow-up
  The composite of 5 clinical endpoints is using a win ratio concept. Mortality has higher priority than Urgent ECMO implantation, urgent heart transplantation or LVAD implantation, unplanned hospitalization for heart failure, improvement of KCCQ by at least 5points, improvement of 6-minute walk test distance by at least 75 meters. Our main approach uses matched pairs of patients. Each pair is 'untied' first on the basis of the most important event (death) and secondly (if necessary) on the lesser event. The numbers of pairs in which the patient on new treatment 'won' and 'lost' are compared to produce the 'win ratio'. The 95% CI and P-value for the win ratio are readily obtained.
Number of unplanned hospitalization for heart failure | Through 24 months when the last subject completes 12 months of follow-up
  The composite of 5 clinical endpoints is using a win ratio concept. Mortality has higher priority than Urgent ECMO implantation, urgent heart transplantation or LVAD implantation, unplanned hospitalization for heart failure, improvement of KCCQ by at least 5points, improvement of 6-minute walk test distance by at least 75 meters. Our main approach uses matched pairs of patients. Each pair is 'untied' first on the basis of the most important event (death) and secondly (if necessary) on the lesser event. The numbers of pairs in which the patient on new treatment 'won' and 'lost' are compared to produce the 'win ratio'. The 95% CI and P-value for the win ratio are readily obtained.
Quality of life assessed by KCCQ score | Through 24 months when the last subject completes 12 months of follow-up
  The composite of 5 clinical endpoints is using a win ratio concept. Mortality has higher priority than Urgent ECMO implantation, urgent heart transplantation or LVAD implantation, unplanned hospitalization for heart failure, improvement of KCCQ by at least 5points, improvement of 6-minute walk test distance by at least 75 meters. Our main approach uses matched pairs of patients. Each pair is 'untied' first on the basis of the most important event (death) and secondly (if necessary) on the lesser event. The numbers of pairs in which the patient on new treatment 'won' and 'lost' are compared to produce the 'win ratio'. The 95% CI and P-value for the win ratio are readily obtained.
Distance in meters at 6-min walking test | Through 24 months when the last subject completes 12 months of follow-up
  The composite of 5 clinical endpoints is using a win ratio concept. Mortality has higher priority than Urgent ECMO implantation, urgent heart transplantation or LVAD implantation, unplanned hospitalization for heart failure, improvement of KCCQ by at least 5points, improvement of 6-minute walk test distance by at least 75 meters. Our main approach uses matched pairs of patients. Each pair is 'untied' first on the basis of the most important event (death) and secondly (if necessary) on the lesser event. The numbers of pairs in which the patient on new treatment 'won' and 'lost' are compared to produce the 'win ratio'. The 95% CI and P-value for the win ratio are readily obtained.

SECONDARY OUTCOMES:
Number of adverse events (AEs) | at 1 month
Number of adverse events (AEs) | at 3 months
Number of adverse events (AEs) | at 6 months
Number of adverse events (AEs) | at 12 months
Number of adverse events (AEs) | at 18 months
Number of adverse events (AEs) | at 24 months
All-cause mortality rate | at 1 month
All-cause mortality rate | at 3 months
All-cause mortality rate | at 6 months
All-cause mortality rate | at 12 months
All-cause mortality rate | at 18 months
All-cause mortality rate | at 24 months
number of ECMO implantation | at 1 month
number of ECMO implantation | at 3 months
number of ECMO implantation | at 6 months
number of ECMO implantation | at 12 months
number of ECMO implantation | at 18 months
number of ECMO implantation | at 24 months
number of urgent heart transplantation | at 1 month
number of urgent heart transplantation | at 3 months
number of urgent heart transplantation | at 12 months
number of urgent heart transplantation | at 18 months
number of urgent heart transplantation | at 24 months
VAD implantation rate | at 1 month
VAD implantation rate | at 3 months
VAD implantation rate | at 6 months
VAD implantation rate | at 12 months
VAD implantation rate | at 18 months
VAD implantation rate | at 24 months
Unplanned hospitalization for heart failure rate | at 1 month
Unplanned hospitalization for heart failure rate | at 3 months
Unplanned hospitalization for heart failure rate | at 6 months
Unplanned hospitalization for heart failure rate | at 12 months
Unplanned hospitalization for heart failure rate | at 18 months
Unplanned hospitalization for heart failure rate | at 24 months
Recurrent hospitalizations rate | at 1 month
  Defined as total number of hospitalizations
Recurrent hospitalizations rate | at 3 months
  Defined as total number of hospitalizations
Recurrent hospitalizations rate | at 6 months
  Defined as total number of hospitalizations
Recurrent hospitalizations rate | at 12 months
  Defined as total number of hospitalizations
Recurrent hospitalizations rate | at 18 months
  Defined as total number of hospitalizations
Recurrent hospitalizations rate | at 24 months
  Defined as total number of hospitalizations
Number of patients with a persistence of the eligibility to LVAD implantation | at 12 and 24 months
  In the GDMT group only
Number of patients with a persistence of the eligibility to LVAD implantation | at 12 months
  In the GDMT group only
Number of days alive out of hospital | at 24 months
New York Heart Association (NYHA) status | at inclusion
New York Heart Association (NYHA) status | at 1 month
New York Heart Association (NYHA) status | at 3 months
New York Heart Association (NYHA) status | at 6 months
New York Heart Association (NYHA) status | at 12 months
New York Heart Association (NYHA) status | at 18 months
New York Heart Association (NYHA) status | at 24 months
Distance in meters at 6-min walking test | at inclusion
Distance in meters at 6-min walking test | at 3 months
Distance in meters at 6-min walking test | at 6 months
Distance in meters at 6-min walking test | at 12 months
Distance in meters at 6-min walking test | at 18 months
Distance in meters at 6-min walking test | at 24 months
Quality of life assessed by European Quality of Life-5 Dimensions (EQ-5D) questionnaire score | at inclusion
Quality of life assessed by European Quality of Life-5 Dimensions (EQ-5D) questionnaire score | at 3 months
Quality of life assessed by European Quality of Life-5 Dimensions (EQ-5D) questionnaire score | at 6 months
Quality of life assessed by European Quality of Life-5 Dimensions (EQ-5D) questionnaire score | at 12 months
Quality of life assessed by European Quality of Life-5 Dimensions (EQ-5D) questionnaire score | at 18 months
Quality of life assessed by European Quality of Life-5 Dimensions (EQ-5D) questionnaire score | at 24 months
Quality of life assessed by KCCQ score | at inclusion
Quality of life assessed by KCCQ score | at 3 months
Quality of life assessed by KCCQ score | at 6 months
Quality of life assessed by KCCQ score | at 12 months
Quality of life assessed by KCCQ score | at 18 months
Quality of life assessed by KCCQ score | at 24 months
Right ventricular function assessed by echocardiographic parameters | at inclusion
Right ventricular function assessed by echocardiographic parameters | at 3 months
Right ventricular function assessed by echocardiographic parameters | at 6 months
Right ventricular function assessed by echocardiographic parameters | at 12 months
Right ventricular function assessed by echocardiographic parameters | at 18 months
Right ventricular function assessed by echocardiographic parameters | at 24 months
Heart failure assessed by N Terminal Pro-Brain Natriuretic Peptide (NT-proBNP) rate | at inclusion
Heart failure assessed by N Terminal Pro-Brain Natriuretic Peptide (NT-proBNP) rate | at 3 months
Heart failure assessed by N Terminal Pro-Brain Natriuretic Peptide (NT-proBNP) rate | at 6 months
Heart failure assessed by N Terminal Pro-Brain Natriuretic Peptide (NT-proBNP) rate | at 12 months
Heart failure assessed by N Terminal Pro-Brain Natriuretic Peptide (NT-proBNP) rate | at 18 months
Heart failure assessed by N Terminal Pro-Brain Natriuretic Peptide (NT-proBNP) rate | at 24 months
Cardio-renal syndrome assessed by rates of Soluble urokinase-type Plasminogen Activator Receptor (SuPAR) | at inclusion
Cardio-renal syndrome assessed by rates of Soluble urokinase-type Plasminogen Activator Receptor (SuPAR) | at 1 month
Cardio-renal syndrome assessed by rates of Soluble urokinase-type Plasminogen Activator Receptor (SuPAR) | at 6 months
Cardio-renal syndrome assessed by rates of Soluble urokinase-type Plasminogen Activator Receptor (SuPAR) | at 12 months
Cardio-renal syndrome assessed by rates of Soluble urokinase-type Plasminogen Activator Receptor (SuPAR) | at 24 months
Cardio-renal syndrome assessed by rates of Interleukin-6 (IL-6) | at inclusion
Cardio-renal syndrome assessed by rates of Interleukin-6 (IL-6) | at 1 month
Cardio-renal syndrome assessed by rates of Interleukin-6 (IL-6) | at 6 months
Cardio-renal syndrome assessed by rates of Interleukin-6 (IL-6) | at 12 months
Cardio-renal syndrome assessed by rates of Interleukin-6 (IL-6) | at 24 months
Cardio-renal syndrome assessed by rates of Kidney Injury Molecule-1 (KIM1) | at inclusion
Cardio-renal syndrome assessed by rates of Kidney Injury Molecule-1 (KIM1) | at 1 month
Cardio-renal syndrome assessed by rates of Kidney Injury Molecule-1 (KIM1) | at 3 months
Cardio-renal syndrome assessed by rates of Kidney Injury Molecule-1 (KIM1) | at 12 months
Cardio-renal syndrome assessed by rates of Kidney Injury Molecule-1 (KIM1) | at 18 months
Cardio-renal syndrome assessed by rates of Kidney Injury Molecule-1 (KIM1) | at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume BAUDRY, Dr, Principal Investigator — CHRU Nancy
Locations (8):
- France (8):
  - CHU Besançon, Besançon
  - Hôpital Pneumologique et Cardiovasculaire Louis Pradel, Bron
  - CHU Caen, Caen
  - La Tronche Hospital / CHU Grenoble, La Tronche
  - Arnaud de Villeneuve Hospital / CHU Montpellier, Montpellier
  - CHU Rouen, Rouen
  - CHU Tours, Tours
  - CHRU, Institut Lorrain du Coeur et des Vaisseaux Louis Mathieu, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No